CLINICAL TRIAL: NCT03424460
Title: Venous Thromboembolism in Myotonic Dystrophy Type 1
Acronym: DM1-VTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: AFM-Téléthon (Funding) (Unknown); Recherche Clinique Paris Descartes Necker Cochin Sainte Anne (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K170601J; 2017-A01634-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2017-12-07; First posted 2018-02-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Myotonic Dystrophy 1
Keywords: Myotonic dystrophy 1; Venous thromboembolism; Pulmonary embolism; Deep vein thrombosis; Hypercoagulability; Thrombophilia; RNA alternative splicing
MeSH Terms: conditions — Myotonic Dystrophy; Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis; Thrombophilia

STUDY DESIGN:
Intervention Model Description: Two populations:
  * Population n°1: prospective, with 3 arms
  * Population n°2: retrospective, with 2 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- population 1-A1 : DM1 with VTE (Experimental): Myotonic dystrophy type 1 patients with a history of venous thromboembolism (pulmonary embolism and/or deep vein thrombosis)
  Interventions: Biological: Haemostasis tests; Biological: Monocytes and megacaryocytes culture and RNA extraction
- population 1-B1 : DM1 without VTE (Active Comparator): Myotonic dystrophy type 1 patients without a history of venous thromboembolism
  Interventions: Biological: Haemostasis tests; Biological: Monocytes and megacaryocytes culture and RNA extraction
- population 1-C1 : Healthy volunteers (Active Comparator): Healthy volunteers without any medical history or treatment
  Interventions: Biological: Haemostasis tests; Biological: Monocytes and megacaryocytes culture and RNA extraction
- population 2-A2 : DM1 liver samples (Experimental): Liver samples of patients with myotonic dystrophy type 1
  Interventions: Genetic: RNA extraction
- population 2-B2 : Healthy liver samples (Active Comparator): Liver samples from patients without any medical history
  Interventions: Genetic: RNA extraction

INTERVENTIONS:
Biological: Haemostasis tests — Venipuncture of 30 milliliters of blood. The following tests will be performed: thromboelastography (TEG®), standard tests of coagulation, genetic thrombophilia, lupus anticoagulant, fibrinolysis markers (Alpha-2-antiplasmin, amidolytic activity, plasmin anti-plasmin complexes, Plasminogen Activator Inhibitor-1 (PAI-1) antigen, plasminogen amydolytic activity), and a global test of fibrinolytic activity.
  Arms: population 1-A1 : DM1 with VTE; population 1-B1 : DM1 without VTE; population 1-C1 : Healthy volunteers
Biological: Monocytes and megacaryocytes culture and RNA extraction — Venipuncture of 60 milliliters of blood. Monocytes and megacaryocytes culture. RNA extraction from monocytes and megacaryocytes.
  Arms: population 1-A1 : DM1 with VTE; population 1-B1 : DM1 without VTE; population 1-C1 : Healthy volunteers
Genetic: RNA extraction — RNA extraction from liver tissue
  Arms: population 2-A2 : DM1 liver samples; population 2-B2 : Healthy liver samples

SUMMARY:
Investigators identified a high risk of deep vein thrombosis and pulmonary embolism in patients presenting myotonic dystrophy type 1 treated in our hospital, 10 times higher than general population matched on age and sex. These venous thromboembolic events were frequently severe and lethal.

Investigators suspect that this high risk of venous thromboembolism is due to coagulation abnormalities specific to myotonic dystrophy type 1.

The purpose of this study is to determine: 1/ if there is a hypercoagulable state in myotonic dystrophy type 1 by testing patient's coagulation, and 2/ if genes encoding factors involved in coagulation have modified expression resulting in this hypercoagulable state.

Understanding the pathophysiology will help preventing venous thromboembolism in these patients.

It is the first study to describe this specific issue.

DETAILED DESCRIPTION:
Investigators have identified in the cohort of 1084 patients presenting myotonic dystrophy type 1 (DM1) a 10% prevalence of venous thromboembolism (VTE) and a 7‰ annual incidence, which is 10-fold higher than in the general population and 3-fold compared to patients with other myopathies.

Patients' clinical presentations were very similar to those observed in patients with severe hypercoagulable states caused by mutations in genes encoding factors involved in coagulation, fibrinolysis or their regulation and represented a frequent cause of death.

To Investigator's knowledge, this association between VTE and DM1 has never been reported to date and no competing project has been initiated on this topic by any other team.

Investigators hypothesize that VTE in DM1 may be related to a hypercoagulable state resulting from an imbalance between coagulation processes and fibrinolysis properties. Because the expression of pathogenic CTG repeats in DM1 leads to a RNA gain-of-function mechanism, Investigators propose these abnormalities may be the consequence of alternative splicing misregulation and/or abnormal gene expression of coagulation, fibrinolysis factors or other factors involved in their regulation.

Investigators applied a candidate gene strategy to screen splicing profiles of 33 genes coding for haemostasis factors in a DM1 context. Using expression large-scale datasets of DM1 tissue samples from skeletal muscle and heart, Investigators identified splicing defects in 4 genes involved in haemostasis, in particular 3 involved in the fibrinolytic system: PLAT, PLAU and SERPINE1. These preliminary analyses were however not performed on liver samples whereas genes coding for haemostasis factors are synthesized and mainly expressed in liver. Analysis of liver and monocytes/megacaryotes RNA samples appears to be an essential step.

The objectives are to (i) study haemostatic properties of a cohort of patients with DM1 with and without personal history of VTE, in order to determine whether a hypercoagulable state may be associated with DM1 and whether it may be correlated to the occurrence of VTE, and (ii) to perform a global transcriptomic approach using massive parallel sequencing (RNAseq) on liver and monocytes/megacaryotes. RNA samples obtained from DM1 patients will help identify candidate genes with altered expression or alternative splicing misregulation that may underlie VTE in DM1.

The study will include two complementary parts in DM1 patients with and without personal history of VTE and healthy volunteers: haemostasis tests, and transcriptomic analysis on RNA samples isolated from liver biopsies and blood monocytes/megacaryocytes samples.Three teams will be involved in the study: Team 1 (clinical study), Team 2 (haematology) and Team 3 (transcriptomic analysis).

Haemostasis tests will be performed by Team 1 and analysed by Team 2 in (i) 100 patients prospectively enrolled in Investigator's Institution by Team 1, aged >18 years, with genetically proven DM1, after providing written informed consent, without any current antithrombotic treatment, including 80 without and 20 with personal history of VTE and (ii) 30 healthy volunteers matched on age and sex. RNAseq will be performed on (i) liver tissue issued from 3 patients with DM1 and 6 controls and (ii) monocytes/megacaryocytes isolated from the blood of 15 patients with DM1 (7 with and 8 without VTE) and 15 controls prospectively enrolled in the study. Inclusion and exclusion criteria will be similar to those of patients included in the study of haemostasis properties.

Liver tissues are already available in a tissue bank. Blood will be prospectively collected in DM1 patients and controls by Team 1. Monocytes and megacaryocytes will be isolated and cultured by Team 2.

Team 3 will extract total RNA from liver samples, monocytes and megacaryocytes to the Centre National de Génotypage for RNA sequencing and perform the analysis of the data and the validation of the newly identified candidates.

The estimated study duration is 72 months, including (i) 66 months for patient inclusions, coagulation testsand monocytes/megacaryocytes isolations, and (ii) 6 months for fibrinolysis tests, RNA extraction and sequencing, data analysis, validation.

Investigators believe the study will have important implications for the clinical management of patients with DM1. Specific strategies will be proposed for the prevention of VTE with potentially larger indications for prophylactic anticoagulant treatments and longer duration after a first episode of VTE.

Regarding the high mortality associated with VTE and the identification in the registry of pulmonary embolism as a frequent cause of death, sudden and non-sudden, in DM1 patients, the modification of these treatment strategies may be associated with an important clinical benefit.The identification of haemostasis abnormalities by coagulation and fibrinolysis tests could be useful for risk stratification in patients with DM1 and could allow targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Population N°1

   * Age over 18 years
   * Patient living in France and with medical insurance
   * Patient having given his informed and written consent
   * DM1 groups: genetically proven DM1
   * VTE groups: at least 1 history of VTE (PE and/or DVT)
   * Healthy volunteers: patient without any medical history (no DM1, no VTE, no thrombophilia), and without taking any anti-thrombotic medication
2. Population N°2

   * Liver tissue of patients with genetically proven DM1 (tissue bank)
   * Liver tissue of patients without DM1 or any history of VTE (tissue bank)

Exclusion Criteria:

* Patient opposed to data collection and analysis

  1. Population N°1
* Genetically proven thrombophilia
* Anti-thrombotic medication
* Hemoglobin levels < 7 g/dL
* Hemoglobin levels < 9 g/dL in case of cardiac of respiratory condition

  2. Population N°2
* Liver tissue quality insufficient for RNA extraction and analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Results of thromboelastography in the 3 arms of population n°1 | 24 months
  Results given in thromboelastography traces

SECONDARY OUTCOMES:
Results of prothrombin time (PT) and activated partial thromboplastin time (APPT) in the 3 arms of population n°1 | 30 months
  Results given in seconds
Results of plasma fibrinogen levels in the 3 arms of population n°1 | 24 months
  Results given in grams per liter
Results of thrombophilia testing in the 3 arms of population n°1 | 24 months
  Testing for:
  * Antithrombin III mutation
  * C protein mutation
  * S protein mutaiton
  * Activated C protein resistance mutation
  * Factor II G20210 mutation
  * Lupus anticoagulant. Results given in: presence or absence (yes or no)
Results of the following fibrinolytic markers: alpha-2-antiplasmine, amidolytic activity, PAI-1 antigen, plasminogen amydolytic activity in the 3 arms of population n°1 | 24 months
  Results given in International Units per milliliters
Results of levels of plasmin anti-plasmin complexes | 24 months
  Results given in picograms per milliliters
Results of global test of fibrinolytic activity by the method of von Kaulla | 24 months
  Results given in hours
Evaluation of coagulation and/or fibrinolysis genes' expression and alternative splicing in the 3 arms of population n°1 and in the 2 arms of population n°2 | 30 months
  Bioanalysis of the patients' transcriptomes after global RNA sequencing, focusing on expression or alternative splicing misregulation of coagulation and/or fibrinolysis genes.
  Results given in : gene name(s) and description

CONTACTS AND LOCATIONS:
Overall Officials: Karim Wahbi, MD, PhD, Principal Investigator — Assistance Publique Hôpitaux de Paris (AP-HP); Denis Duboc, MD, PhD, Study Director — Assistance Publique Hôpitaux de Paris (AP-HP); Michaela Fontenay, MD, PhD, Study Chair — Assistance Publique Hôpitaux de Paris (AP-HP); Denis Furling, Md, PhD, Principal Investigator — Université Paris 6 Pierre et Marie Curie
Locations (1):
- Service de Cardiologie - Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Udd B, Krahe R. The myotonic dystrophies: molecular, clinical, and therapeutic challenges. Lancet Neurol. 2012 Oct;11(10):891-905. doi: 10.1016/S1474-4422(12)70204-1. PMID 22995693
- [Background] Mathieu J, De Braekeleer M, Prevost C. Genealogical reconstruction of myotonic dystrophy in the Saguenay-Lac-Saint-Jean area (Quebec, Canada). Neurology. 1990 May;40(5):839-42. doi: 10.1212/wnl.40.5.839. PMID 2330114
- [Background] Fu YH, Pizzuti A, Fenwick RG Jr, King J, Rajnarayan S, Dunne PW, Dubel J, Nasser GA, Ashizawa T, de Jong P, et al. An unstable triplet repeat in a gene related to myotonic muscular dystrophy. Science. 1992 Mar 6;255(5049):1256-8. doi: 10.1126/science.1546326.
- [Background] Mahadevan M, Tsilfidis C, Sabourin L, Shutler G, Amemiya C, Jansen G, Neville C, Narang M, Barcelo J, O'Hoy K, et al. Myotonic dystrophy mutation: an unstable CTG repeat in the 3' untranslated region of the gene. Science. 1992 Mar 6;255(5049):1253-5. doi: 10.1126/science.1546325.
- [Background] Brook JD, McCurrach ME, Harley HG, Buckler AJ, Church D, Aburatani H, Hunter K, Stanton VP, Thirion JP, Hudson T, et al. Molecular basis of myotonic dystrophy: expansion of a trinucleotide (CTG) repeat at the 3' end of a transcript encoding a protein kinase family member. Cell. 1992 Feb 21;68(4):799-808. doi: 10.1016/0092-8674(92)90154-5. PMID 1310900
- [Background] Day JW, Ranum LP. RNA pathogenesis of the myotonic dystrophies. Neuromuscul Disord. 2005 Jan;15(1):5-16. doi: 10.1016/j.nmd.2004.09.012. Epub 2004 Nov 26. PMID 15639115
- [Background] Mankodi A, Logigian E, Callahan L, McClain C, White R, Henderson D, Krym M, Thornton CA. Myotonic dystrophy in transgenic mice expressing an expanded CUG repeat. Science. 2000 Sep 8;289(5485):1769-73. doi: 10.1126/science.289.5485.1769. PMID 10976074
- [Background] Tian B, White RJ, Xia T, Welle S, Turner DH, Mathews MB, Thornton CA. Expanded CUG repeat RNAs form hairpins that activate the double-stranded RNA-dependent protein kinase PKR. RNA. 2000 Jan;6(1):79-87. doi: 10.1017/s1355838200991544. PMID 10668800
- [Background] Charizanis K, Lee KY, Batra R, Goodwin M, Zhang C, Yuan Y, Shiue L, Cline M, Scotti MM, Xia G, Kumar A, Ashizawa T, Clark HB, Kimura T, Takahashi MP, Fujimura H, Jinnai K, Yoshikawa H, Gomes-Pereira M, Gourdon G, Sakai N, Nishino S, Foster TC, Ares M Jr, Darnell RB, Swanson MS. Muscleblind-like 2-mediated alternative splicing in the developing brain and dysregulation in myotonic dystrophy. Neuron. 2012 Aug 9;75(3):437-50. doi: 10.1016/j.neuron.2012.05.029. PMID 22884328
- [Background] Nakamori M, Sobczak K, Puwanant A, Welle S, Eichinger K, Pandya S, Dekdebrun J, Heatwole CR, McDermott MP, Chen T, Cline M, Tawil R, Osborne RJ, Wheeler TM, Swanson MS, Moxley RT 3rd, Thornton CA. Splicing biomarkers of disease severity in myotonic dystrophy. Ann Neurol. 2013 Dec;74(6):862-72. doi: 10.1002/ana.23992. PMID 23929620
- [Background] Mankodi A, Takahashi MP, Jiang H, Beck CL, Bowers WJ, Moxley RT, Cannon SC, Thornton CA. Expanded CUG repeats trigger aberrant splicing of ClC-1 chloride channel pre-mRNA and hyperexcitability of skeletal muscle in myotonic dystrophy. Mol Cell. 2002 Jul;10(1):35-44. doi: 10.1016/s1097-2765(02)00563-4. PMID 12150905
- [Background] Fugier C, Klein AF, Hammer C, Vassilopoulos S, Ivarsson Y, Toussaint A, Tosch V, Vignaud A, Ferry A, Messaddeq N, Kokunai Y, Tsuburaya R, de la Grange P, Dembele D, Francois V, Precigout G, Boulade-Ladame C, Hummel MC, Lopez de Munain A, Sergeant N, Laquerriere A, Thibault C, Deryckere F, Auboeuf D, Garcia L, Zimmermann P, Udd B, Schoser B, Takahashi MP, Nishino I, Bassez G, Laporte J, Furling D, Charlet-Berguerand N. Misregulated alternative splicing of BIN1 is associated with T tubule alterations and muscle weakness in myotonic dystrophy. Nat Med. 2011 Jun;17(6):720-5. doi: 10.1038/nm.2374. Epub 2011 May 29. PMID 21623381
- [Background] Rau F, Laine J, Ramanoudjame L, Ferry A, Arandel L, Delalande O, Jollet A, Dingli F, Lee KY, Peccate C, Lorain S, Kabashi E, Athanasopoulos T, Koo T, Loew D, Swanson MS, Le Rumeur E, Dickson G, Allamand V, Marie J, Furling D. Abnormal splicing switch of DMD's penultimate exon compromises muscle fibre maintenance in myotonic dystrophy. Nat Commun. 2015 May 28;6:7205. doi: 10.1038/ncomms8205. PMID 26018658
- [Background] Savkur RS, Philips AV, Cooper TA. Aberrant regulation of insulin receptor alternative splicing is associated with insulin resistance in myotonic dystrophy. Nat Genet. 2001 Sep;29(1):40-7. doi: 10.1038/ng704. PMID 11528389
- [Background] Yadava RS, Frenzel-McCardell CD, Yu Q, Srinivasan V, Tucker AL, Puymirat J, Thornton CA, Prall OW, Harvey RP, Mahadevan MS. RNA toxicity in myotonic muscular dystrophy induces NKX2-5 expression. Nat Genet. 2008 Jan;40(1):61-8. doi: 10.1038/ng.2007.28. Epub 2007 Dec 16. PMID 18084293
- [Background] Kearon C. Natural history of venous thromboembolism. Circulation. 2003 Jun 17;107(23 Suppl 1):I22-30. doi: 10.1161/01.CIR.0000078464.82671.78. PMID 12814982
- [Background] Torbicki A, Perrier A, Konstantinides S, Agnelli G, Galie N, Pruszczyk P, Bengel F, Brady AJ, Ferreira D, Janssens U, Klepetko W, Mayer E, Remy-Jardin M, Bassand JP; ESC Committee for Practice Guidelines (CPG). Guidelines on the diagnosis and management of acute pulmonary embolism: the Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). Eur Heart J. 2008 Sep;29(18):2276-315. doi: 10.1093/eurheartj/ehn310. Epub 2008 Aug 30. PMID 18757870
- [Background] Goldhaber SZ, Visani L, De Rosa M. Acute pulmonary embolism: clinical outcomes in the International Cooperative Pulmonary Embolism Registry (ICOPER). Lancet. 1999 Apr 24;353(9162):1386-9. doi: 10.1016/s0140-6736(98)07534-5. PMID 10227218
- [Background] Karwinski B, Svendsen E. Comparison of clinical and postmortem diagnosis of pulmonary embolism. J Clin Pathol. 1989 Feb;42(2):135-9. doi: 10.1136/jcp.42.2.135. PMID 2921354
- [Background] Dalen JE. Pulmonary embolism: what have we learned since Virchow? Natural history, pathophysiology, and diagnosis. Chest. 2002 Oct;122(4):1440-56. doi: 10.1378/chest.122.4.1440. No abstract available. PMID 12377877
- [Background] Anderson FA Jr, Spencer FA. Risk factors for venous thromboembolism. Circulation. 2003 Jun 17;107(23 Suppl 1):I9-16. doi: 10.1161/01.CIR.0000078469.07362.E6. PMID 12814980
- [Background] Goldhaber SZ. Risk factors for venous thromboembolism. J Am Coll Cardiol. 2010 Jun 29;56(1):1-7. doi: 10.1016/j.jacc.2010.01.057. PMID 20620709
- [Background] Oger E. Incidence of venous thromboembolism: a community-based study in Western France. EPI-GETBP Study Group. Groupe d'Etude de la Thrombose de Bretagne Occidentale. Thromb Haemost. 2000 May;83(5):657-60. PMID 10823257
- [Background] Achiron A, Barak Y, Magal N, Shohat M, Cohen M, Barar R, Gadoth N. Abnormal liver test results in myotonic dystrophy. J Clin Gastroenterol. 1998 Jun;26(4):292-5. doi: 10.1097/00004836-199806000-00016. PMID 9649014
- [Background] Wang ET, Cody NA, Jog S, Biancolella M, Wang TT, Treacy DJ, Luo S, Schroth GP, Housman DE, Reddy S, Lecuyer E, Burge CB. Transcriptome-wide regulation of pre-mRNA splicing and mRNA localization by muscleblind proteins. Cell. 2012 Aug 17;150(4):710-24. doi: 10.1016/j.cell.2012.06.041. PMID 22901804
- [Background] Batra R, Charizanis K, Manchanda M, Mohan A, Li M, Finn DJ, Goodwin M, Zhang C, Sobczak K, Thornton CA, Swanson MS. Loss of MBNL leads to disruption of developmentally regulated alternative polyadenylation in RNA-mediated disease. Mol Cell. 2014 Oct 23;56(2):311-322. doi: 10.1016/j.molcel.2014.08.027. Epub 2014 Sep 25. PMID 25263597